CLINICAL TRIAL: NCT04784052
Title: TCRαβ+ T-cell/CD19+ B-cell Depleted Hematopoietic Grafts and a Reduced Intensity Preparative Conditioning Regimen Containing JSP191 (Briquilimab) to Achieve Engraftment and Blood Reconstitution in Patients With Fanconi Anemia
Brief Title: Depleted Donor Stem Cell Transplant in Children and Adults With Fanconi Anemia After Being Conditioned With a Regimen Containing Briquilimab
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Porteus, Matthew, MD (Other)
Responsible Party: Principal Investigator, Rajni Agarwal, Associate Professor of Pediatrics, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-60108
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Fanconi Anemia
Keywords: Cell Transplants; Grafts; Stem Cells
MeSH Terms: conditions — Fanconi Anemia | interventions — Cyclophosphamide; fludarabine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Depleted Stem Cell Transplant with JSP-191 Conditioning (Experimental): Participants will receive an infusion of donor stem cells which have been depleted of αβ+T cells using the CliniMACS System device. Before the stem cell transplant, they will receive a reduced-intensity preparative regimen containing JSP191 in combination with rATG, cyclophosphamide, fludarabine and rituximab.
  Interventions: Drug: JSP191; Device: CliniMACS Prodigy System; Biological: Depleted Stem Cell Transplant; Biological: Rabbit Anti-Thymoglobulin (rATG); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab
- Depleted Stem Cell Transplant without JSP-191 Conditioning (Experimental): Participants will receive an infusion of donor stem cells which have been depleted of αβ+T cells using the CliniMACS System device. Before the stem cell transplant, they will receive a reduced-intensity preparative regimen containing rATG, cyclophosphamide, fludarabine and rituximab.
  Interventions: Device: CliniMACS Prodigy System; Biological: Depleted Stem Cell Transplant; Biological: Rabbit Anti-Thymoglobulin (rATG); Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: JSP191 — Participants will receive a single IV dose at start of conditioning
  Arms: Depleted Stem Cell Transplant with JSP-191 Conditioning
Device: CliniMACS Prodigy System — The device used to remove the αβ+T cells from donor stem cell transplant before being given to the recipient
Biological: Depleted Stem Cell Transplant — TCRαβ+ T-cell/CD19+ B-cell depleted hematopoietic cells will be administered by IV after completion of conditioning regimen.
Biological: Rabbit Anti-Thymoglobulin (rATG) — 3 consecutive daily doses of rATG will be given by IV during conditioning
Drug: Cyclophosphamide — 4 consecutive daily doses of cyclophosphamid will be given by IV during conditioning
  Other Names: Cytoxan
Drug: Fludarabine — 4 consecutive daily doses of fludarabine will be given by IV during conditioning
Drug: Rituximab — 1 dose of rituximab will be given at the end of conditioning

SUMMARY:
The objective of this clinical trial is to develop a cell therapy for Fanconi Anemia which enables enhanced donor hematopoietic and immune reconstitution with decreased toxicity by transplanting depleted stem cells from a donor with and without using an experimental antibody treatment called JSP-191 as a part of conditioning. This experimental treatment will hopefully cause fewer side effects than chemotherapy (the current standard of care method).

Participants will be administered the conditioning regimen, are assessed until they receive the depleted stem cell infusion, and will be followed for up to 2 years after the cell infusion.

ELIGIBILITY:
Inclusion Criteria:

All patients must have:

1. Fanconi Anemia diagnosis as demonstrated by abnormal chromosome breakage studies with increased sensitivity to mitomycin-C (MMC) or diepoxybutane (DEB) and at least one mutation in a known Fanconi-associated gene
2. Bone marrow failure (defined by reduction in at least one cell line on two separate occasions at least one month apart (e.g., platelet count of <100,000 per cubic millimeter, hemoglobin <9 gm/dl and/or absolute neutrophil count (ANC) of <1000/mm)
3. Age of ≥2 years
4. Consenting ≥5/10 HLA-matched related or unrelated donor available for apheresis
5. Organ function defined as:

   1. Serum Creatinine <2.0 mg/dL and corrected creatinine clearance/cystatin cL >60 mL/min/1.73m^2 without dialysis
   2. Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and diffusing capacity of the lung for carbon monoxide (DLCO) corrected for hemoglobin and volume, >50% predicted by pulmonary function tests (PFTs)
   3. For patients unable to cooperate for PFTs, criteria are no evidence of dyspnea at rest, no exercise intolerance, and no requirement for supplemental oxygen with spO2 >93%
   4. Shortening fraction of ≥29% or ejection fraction of ≥45% by echocardiogram
   5. Serum total bilirubin of <4 x ULN
   6. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5 x ULN
   7. Prothrombin time international normalized ratio (PT INR) and partial thromboplastin time (PTT) <1.5 x ULN
6. Life expectancy of at least 2 years
7. Patients of childbearing potential must be willing to use an effective contraceptive method for the duration of the peri-transplant conditioning through hematopoietic recovery
8. Patients and/or parents or legal guardians must be able to provide written informed consent and authorize use and disclosure of personal health information in accordance with Health Insurance Portability and Accountability Act

Exclusion Criteria:

1. Patients with available and consenting 10/10 HLA-identical sibling donor for apheresis
2. Patients with any acute or uncontrolled infections at the time of enrollment, including bacterial, fungal or viral
3. Patients who are seropositive for HIV-I/II or HTLV-I/II.
4. Patients receiving any other investigational agents or other biological, chemotherapy, or radiation therapy within 14 days of enrollment
5. Patients with any active malignancies, myelodysplastic syndrome or other concerns for high-risk bone marrow disease
6. Patients who received androgens in last 3 months
7. Pregnant or lactating women
8. Women who are nursing and do not wish to discontinue breastfeeding
9. Lansky/Karnofsky performance score <50%.
10. Any other medical condition or history that, in the opinion of the Principal Investigator, could pose a significant safety risk to the participant or jeopardize the integrity of the study
11. Patients who, in the opinion of the Principal Investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants without grade 3 and 4 treatment-emergent adverse events (TEAEs) (infusion related reactions). | From start of conditioning regimen administration until cell infusion (up to 30 days)
  Recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Number of participants without grade 3 and 4 treatment-emergent adverse events (TEAEs) (infusion related reactions) following infusion of TCRαβ+ T-cell/CD19+ B-cell depleted hematopoietic graft transplantation | Up to 2 years post-cell infusion
Number of participants able to achieve donor engraftment | Assessed at Day +42 post-cell infusion
  Participants have achieved engraftment when absolute Neutrophil Count (ANC) is above 500/mm^3 for three consecutive laboratory values obtained on different days post cell transplantation with >1% CD15 donor chimerism
Number of participants who are able to have donor engraftment persist at the same rate or better compared to alternative hematopoietic cell transplant regimens for this patient population | Assessed at Day +100 post-cell infusion

SECONDARY OUTCOMES:
Serum concentration of JSP191 | Prior to start of conditioning regimen, and 5 minutes, 4 hours, +2, +3, +4, +6, +8, +10 days after start of conditioning regimen, and day of cell infusion
  Assessed as serum concentrations in the peripheral blood from administration until time of cell infusion
Serum concentration of rATG | Prior to start of rATG infusion; 15 minutes after first, second, and third rATG infusion; day of cell infusion; and week +1, week +2 and week +12 post cell infusion
  Assessed as serum concentrations in the peripheral blood from administration until time of cell infusion
Serum concentration of fludarabine | Prior to start of fludarabine infusion, and 15 minutes, 1 hour, 3 hours, and 6 hours after the fludarabine infusion
  Assessed as serum concentrations in the peripheral blood from administration until time of cell infusion
Participants who do not develop mucositis | Start of conditioning regimen until +12 weeks post-cell infusion (up to 15 weeks)
  Mucositis incidence will be scored using the CTC criteria
Participants who do not develop veno-occlusive disease (VOD) | Start of conditioning regimen until +12 weeks post-cell infusion (up to 15 weeks)
  VOD incidence will be scored using the Modified Seattle criteria
Number of participants who achieve hematopoietic recovery | Up to 107 weeks (after start of conditioning regimen through Week +104 post-cell infusion)
  Hematopoietic recovery defined by hemoglobin >8g/dL and platelets >20k/dL without transfusion support achieved on 7 days post-graft transplantation documented on hematologic monitoring
Number of participants who achieve donor engraftment | Weeks +1 through +104 post-cell infusion
  Engraftment measured as peripheral blood (total, CD15+, CD3+, CD19+, CD56+, and CD34+) and bone marrow (total and CD34+) chimerism by STR analysis
Number of participants who achieve immunologic recovery | Weeks +1 through +104 post-cell infusion
  Immunologic recovery defined as >200/uL CD3+ T-cells and as assessed by percent and absolute numbers of T (CD3), B (CD19) and NK (CD56) cells by CBC differential studies and flow cytometry for lymphocyte lineages
Number of participants who develop Grade I-IV acute graft-vs-host disease (GvHD) | Day +100 post-cell infusion
Number of participants who develop chronic graft-vs-host disease (GvHD) | Day +100 through Week +104 post-cell infusion
Number of participants who achieve disease-free survival | Up to 104 weeks (from time of cell infusion through Week +104)
  Disease-free defined by improved DEB-induced chromosomal breakage analysis in peripheral blood lymphocyte cultures

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Agarwal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal R, Bertaina A, Soco C, Long-Boyle JR, Saini G, Kunte N, Hiroshima L, Chan YY, Willner H, Krampf MR, Nofal R, Barbarito G, Sen S, Van Hentenryck M, Walck E, Scheck A, Perriman RJ, Bouge A, Istomina E, Din HN, Klinger EF, Cheng JC, Wlodarski MW, Boelens JJ, Shizuru JA, Pang WW, Weinberg K, Parkman R, Roncarolo MG, Porteus M, Czechowicz A. Irradiation- and busulfan-free stem cell transplantation in Fanconi anemia using an anti-CD117 antibody: a phase 1b trial. Nat Med. 2025 Sep;31(9):3183-3190. doi: 10.1038/s41591-025-03817-1. Epub 2025 Jul 22. PMID 40696207